CLINICAL TRIAL: NCT01653366
Title: Effect of a Goal Setting Intervention on Exercise in Women With Metastatic Breast Cancer: An Exploration of The Lipogenic Pathway
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: primary goal not achievable
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D11282
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A-Pedometer and Goal setting (Experimental): Physical Activity Goal Setting
  Patients receive physical therapy (PT) consult, educational materials, and telephone calls and are contacted weekly/monthly for physical activity (PA) goal setting with registered nurse (RN). Physical Activity completed is measured with pedometers and recorded on patient log.
  Interventions: Behavioral: Physical Activity Goal Setting
- ARM B (No Intervention): Patients receive standard physical activity recommendations and follow up.

INTERVENTIONS:
Behavioral: Physical Activity Goal Setting — Will include an initial physical therapy (PTA) consult to set exercise goals to increase physical activity by 6000 steps per week over the course of the trial, viewing of the "Exercise and Breast Cancer" digital video disc (DVD, followed by 10 regular phone calls or RN visits (weekly for the first month, then monthly) to follow up on whether or not those goals are being met and, if not, how best to meet them.
  Arms: Arm A-Pedometer and Goal setting

SUMMARY:
This study is a randomized prospective clinical trial of women with metastatic breast cancer. The purpose of the study is to test if an intervention of regular physical activity review and physical activity goal setting will allow the subjects to achieve a moderate increase in physical activity of 6,000 steps per week. The physical activity review will consist of weekly telephone call to inquire about symptoms and to set physical activity goals. The study will also look to see if the goal setting intervention will affect the time to progression, change in BMI, and quality of life. Quality of life will be measured by answers to questionnaires provided to subjects at regular intervals during the course of the study. Finally, the study will examine the impact of physical activity on expression of tumor molecular molecules, insulin levels, and estradiol levels.

Through an intervention of regular physical activity review and goal setting, the investigators hypothesize that a moderate increase in level of physical activity of 6000 steps per week or more can be obtained by patients with metastatic breast cancer who receive a goal setting intervention. The investigators propose that those who are able to achieve and maintain greater than or equal to 22500 steps per week will demonstrate biologic and molecular differences compared to those who are not able to achieve that level of physical activity. The investigators expect that people who are more active will have longer to progression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with measurable per Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 and biopsy-able (as determined by Co-Investigator John Gemery, MD) metastatic carcinoma of the breast.
* Physically able to undertake a moderate physical activity program.
* Greater than 4 weeks from any radiation treatments for metastatic disease.
* standard of care biopsy must occur within 30 days of registration.
* Able to follow directions and fill out questionnaires and physical activity diaries in English.
* Willing to consent to biopsies and be randomly assigned to one of two study arms which may or may not include physical activity goal setting.
* Consents to be contacted via phone or internet (see Appendix K).
* No to all questions on Physical Activity Readiness Questionnaire (see appendix A) or approved by primary oncologist or other care provider provider for participation.
* Hb >10 without transfusion, liver function tests less than 3 times upper limits of normal, normal thyroid-stimulating hormone (TSH), absolute neutrophil count (ANC) >1500.
* Karnofsky performance status ≥ 80%
* Previous Physical Therapy consultation and treatments acceptable.
* Participation in other trials acceptable.
* CNS disease that is treated and stable by MRI for at least 6 months

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients unable to give informed consent indicating they are aware of the investigational nature of this treatment, prior to entry into the study.
* Pregnant or nursing women.
* Patients with any untreated (CNS) disease.
* Patients with other active cancers requiring treatment.
* Patients with clotting or bleeding disorder precluding biopsy.
* Patients with significant cardiovascular disease, including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months or serious cardiac arrhythmias will be excluded.
* Current use of supplements containing conjugated linoleic acid, or use within the 30 days preceding registration.
* Persons with a known diagnosis of diabetes are not eligible. Prior use of metformin allowable if previously enrolled on MA.32 trial as part of their adjuvant therapy for early stage breast cancer.
* Persons of male gender.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as a result of a goal setting intervention using pedometer data and exercise logs. | Baseline, 2 month, 3 month, 4 month, 5 month, 6 months
  To increase physical activity levels by at least 6000 steps/wk over 6 months using a goal setting intervention

SECONDARY OUTCOMES:
Secondary objectives: Time to progression | baseline, 6 months
  goal-setting intervention versus standard of care: Time to progression
Change in Body Mass Index (BMI) | Baseline, 2 month, 3 month, 4 month, 5 month, 6 months
Health related quality of life | baseline, 6 months
  As measured by questionnaires: FACIT-F and diet survey
Correlative Science outcomes in peripheral blood | baseline, 6 months
  serum estradiol and fasting insulin levels
Correlative science outcomes in tissue biopsies | baseline, 6 months
  relative protein expression of Lipoprotein Lipase (LPL), Cluster of Differentiation 36 (CD36), Spot 14 and fatty acid synthase (FASN) of the original tumor to the metastatic tumor at baseline and at the end of the study.
correlative science in >= 22500 steps | baseline, 6 months
  Compare correlative science outcomes in those who achieve greater than or equal to 22500 steps/ week to those who do not.
participants who achieve >= 22500 steps/week | 6 months
  Determine the proportion of participants who are able to achieve greater than or equal to 22,500 steps/week

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States